CLINICAL TRIAL: NCT01087892
Title: Probiotics in Preventing Antibiotic Associated Diarrhoea Including Clostridium Difficile Infection
Acronym: NU278
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sussex (Other)
Collaborators: Danone Institute International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UKCRN7582
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Diarrhoea; Clostridium Difficile
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary supplement Probiotic drink (Active Comparator): Double blind
  Probiotic containing the live strain 100g/day orally, twice daily for the duration of the course of antibiotics plus seven days
  Interventions: Dietary Supplement: Probiotic drink containing the live strain
- Dietary supplement probiotic placebo drink (Placebo Comparator): Double blind
  'placebo' is actually a control product
  Placebo drink contains no strain 100gs orally, twice daily for the duration of the course of antibiotics plus seven days
  Interventions: Dietary Supplement: placebo probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic drink containing the live strain — Probiotic drink contains no strain
  Arms: Dietary supplement Probiotic drink
Dietary Supplement: placebo probiotic — Placebo product is a sweetened flavoured, non fermented, acidified dairy drink
  Arms: Dietary supplement probiotic placebo drink

SUMMARY:
Antibiotics are currently required to treat patients in hospital when they have an infection, but these antibiotics can cause side effects such as diarrhoea and in some patients a serious form of gut infection with an organism called Clostridium difficile. This organism can produce toxins in the gut causing a severe form of diarrhoea associated with a lot of ill health, and in some circumstances can be fatal. Some studies have shown that yogurts' or Probiotics' (special drinks with a defined concentration of useful bacteria) taken by patients can have a beneficial effect in reducing the diarrhoea associated with antibiotics use. The aim of the present study is to find out whether the use of one of these Probiotics in hospitalised patients taking antibiotics will result in less diarrhoea, less Clostridium difficile infection, as well as cost saving. The study will also analyze the effects of probiotics on quality of life and length of hospital stay.

DETAILED DESCRIPTION:
As part of this study, we will look at both microbiological and immunological markers, in addition to analyzing the overall cost implications by analysis of health economics.

ELIGIBILITY:
Inclusion Criteria:

* Male/female patients, above 55 years of age Patient has given written informed consent/Assent to take part in the study Patients are receiving antibiotics as inpatients Patients prescribed therapy with single or multiple antibiotics (oral or IV) will be included Antibiotic therapy must be indicated for a minimum of 72 hours Patients must be able to take medication orally Inclusion in the study is approved by the admitting consultant and validated by a member of the trial team within 48 hours

Exclusion Criteria:

* Age less than 55 years Pregnancy Patients on PEG feed. Diarrhoea on admission or within the preceding week Severe life-threatening illness

Subjects with allergy or hypersensitivity to any component of the study product (e.g.: allergy or hypersensitivity to milk proteins) Subjects who had any surgery or intervention in the last 4 weeks Subjects enrolled in another clinical study in the last 4 weeks Subjects who are thought not to comply with the clinical study Subjects presenting with a severe evolving or active pathology or infection of the gastrointestinal tract such as inflammatory bowel disease, Crohn's disease or ulcerative colitis, diverticular disease or liver cirrhosis.

Any condition affecting the pancreas including acute and chronic pancreatitis Patients who had a surgical operation in their bowels in the preceding 3 months A medical condition such that the life expectancy of the patient is predicted at less than 3 months by the admitting consultant and validated by a member of the trial team Immune-suppressed patients (e.g. HIV) Steroid use of Prednisolone greater than 10mg a day (or equivalent of Dexamethasone) for over 2 weeks prior to entering the trial Patients on Cytotoxic drugs Post-transplant patients Any clinical condition affecting the pancreas including acute and chronic pancreatitis Patients with prosthetic heart valves or a history of endocarditis. Patients who have taken probiotic drinks containing live organisms or over the counter probiotic preparations in the past seven days (see Appendix 10) Foreign travel in the last 7 days

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1126 (Actual)
Dates: Start 2009-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The incidence of diarrhoea | regular intervals for 28days from entry to trial
  The incidence of antibiotic associated diarrhoea in the active and placebo group by the end of the follow up period

SECONDARY OUTCOMES:
incidence and duration of Clostridium difficile toxin | regular intervals for 28 days from entry to trial
  The incidence and duration of Clostridium difficile toxin detected by ELISA positive testing from a stool sample taken at the onset of diarrhoea in the active and placebo groups
The rate of recurrence of antibiotic associated diarrhoea in the active and placebo groups to the end of the follow up period | regular intervals for 28 days from entry to trial
  The rate of recurrence of antibiotic associated diarrhoea in the active and placebo groups to the end of the follow up period
rate of recurrence of Clostridium difficile toxin positive diarrhoea | regular intervals for 28 days from entry to trial
  The rate of recurrence of Clostridium difficile toxin positive diarrhoea in the active and placebo groups from hospital discharge until the end of the follow-up period
The quality of life in the active and placebo groups at enrollment into the study | regular intervals for 28 days from entry to trial
The length of hospital stay from enrollment into the study until the end of the follow up period in the active and placebo groups The cost-effectiveness as evidenced by health economic calculations | regular intervals for 28 days from entry to trial

CONTACTS AND LOCATIONS:
Overall Officials: Chakravarthi Rajkumar, Study Chair — University of Sussex
Locations (26):
- United Kingdom (26):
  - Ashford and St Peters Hospital, Ashford
  - Blackpool Vicotria Hospital, Blackpool
  - Royal Sussex County Hospital, Brighton
  - Cambridge University Hospital Trust, Cambridge
  - Broomfield Hospital, Chelmsford
  - St.Richards Hospital, Chichester
  - Colchester Hospitals University, Colchester
  - Ealing Hospital, Ealing
  - Eastbourne District General Hospital, Eastbourne
  - Frimley Park Hospital, Frimley
  - Princess Royal Hospital, Haywards Heath
  - Hillingdon Hospital, Hillingdon
  - Lancashire Teaching Hospital, Lancaster
  - University Hosppitals of Leicester, Leicester
  - Lewisham Helathcare NHS Trust, Lewisham
  - Kings College Hospital, London
  - St Georges Hospital London, London
  - Queen Elizabeth Queen Mother Hospital, Margate
  - University Hospitals of Morecambe Bay, Morecambe
  - Norfolk and Norwich University, Norwich
  - Portsmouth Hospitals NHS Trust, Portsmouth
  - Worcestershire Acute Hospitals, Redditch
  - East Surrey Hospital, Redhill
  - Maidstone and Tunbridge Wells NHS Trust, Royal Tunbridge Wells
  - University Hospital Southampton, Southampton
  - Yeovil District Hospital, Yeovil